CLINICAL TRIAL: NCT01414010
Title: Effects of Mushroom Extract, S Boulardii and Amoxicillin on the Human Microbiome
Brief Title: Effects of Pre-, Pro- & Anti-biotics on Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Hong Kong Association for Health Care (Unknown); Integrated Chinese Medicine Holdings (Unknown)
Responsible Party: Principal Investigator, Ciaran Kelly, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010P000319
Record Dates: First submitted 2011-08-05; First posted 2011-08-11 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Human Gut Microbiota
Keywords: healthy volunteers; gut microbiota; gut microbiome; prebiotic; probiotic; antibiotic; antibiotic-associated diarrhea; intestinal bacterial overgrowth
MeSH Terms: interventions — VPS Coriolus versicolor extract; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Prebiotic (Active Comparator)
  Interventions: Dietary Supplement: Trametes versicolor extract
- Probiotic (Active Comparator)
  Interventions: Dietary Supplement: Saccharomyces boulardii
- Antibiotic (Active Comparator)
  Interventions: Drug: Amoxicillin
- Control (No Intervention): Control group, no intervention given.

INTERVENTIONS:
Dietary Supplement: Trametes versicolor extract — 1,200 mg, 3 times daily on an empty stomach for 14 days
  Other Names: turkey tail
  Arms: Prebiotic
Dietary Supplement: Saccharomyces boulardii — 250 mg, 3 times daily on an empty stomach for 14 days
  Arms: Probiotic
Drug: Amoxicillin — 250 mg 3 times daily at least 1 hour before meals for 7 days
  Arms: Antibiotic

SUMMARY:
The purpose of this study is to compare and contrast the effects of a prebiotic (Trametes Versicolor), a probiotic (Saccharomyces boulardii) and an antibiotic (amoxicillin) on the gut microbiota of healthy volunteers. It is expected that treatment will result in the rapid and reproducible alterations in fecal microbiota that will spontaneously reverse in the weeks after treatment is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 39 years (male or female)
* Good general health
* Able to comply with study requirements and to provide informed consent
* For women of childbearing potential
* A negative urine pregnancy test immediately prior to starting the study treatment
* Agreement to comply with approved methods of contraception during the period of active study treatment (not required during follow-up)

Exclusion Criteria:

* Any diagnosed autoimmune disease
* History of organ transplantation
* Known chronic or recurrent systemic disorder associated with immunocompromise
* A history of allergy or hypersensitivity to mushroom or mushroom extract, brewer's or baker's yeast or to penicillins or cephalosporins (including amoxicillin).
* History of severe allergic reaction (requiring hospital admission and/or the administration of parenteral medication or associated with dyspnoea, wheezing, hypotension, loss of consciousness).
* Systemic antibacterial therapy during the 3 months prior to study enrollment
* New prescription medications during the 4 weeks prior to study enrollment
* Prescription or OTC medications or supplements that are known to alter gut function or microflora (i.e. acid antisecretory drugs, probiotics) during the 4 weeks prior to study enrollment
* Active gastrointestinal or metabolic disease
* Prior gastrointestinal surgery (apart from appendectomy or cholecystectomy)
* History of chronic constipation with passage of fewer than 3 spontaneous bowel movements per week on average or chronic or recurrent diarrhea with spontaneous bowel movements more often than 3 times daily
* Any condition or personal circumstance that, in the opinion of the investigator, renders the subject unlikely or unable to comply with the full study protocol.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran P Kelly, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prebiotic | Probiotic | Antibiotic | Control
Started | 8 | 8 | 8 | 8
Completed | 6 | 8 | 8 | 8
Not Completed | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prebiotic | Probiotic | Antibiotic | Control | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (13.7) | 32.9 (9.8) | 32.1 (8.9) | 29.9 (10.3) | 32 (10.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 5 | 22
  Male | 3 | 2 | 2 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Bacteria Prevalence in Stool
Description: The most prevalent bacterial genera within the study population
  Before Treatment: Average of Day -7 and Day 0 During Treatment: Average of Days 10 and 14 After Treatment: Average of Days 21, 28, and 56
Time Frame: Day 0 to 56
Population: The investigators expanded their studies on the probiotic (Saccharomyces boulardii) to constitute a full, separate study. Reference: NCT01473368.
Measure: Mean (Standard Deviation); unit: percentage of bacterial genera in stool
Groups:
- Amoxicillin - Before Treatment; Amoxicillin - During Treatment; Amoxicillin - After Treatment: Amoxicillin: 250 mg 3 times daily at least 1 hour before meals for 7 days
- Control: Control group - no intervention given.
- Trametes Versicolor Extract - Before Treatment; Trametes Versicolor Extract - During Treatment; Trametes Versicolor Extract - After Treatment: Trametes versicolor extract: 1,200 mg, 3 times daily on an empty stomach for 14 days
- Saccharomyces Boulardii - Before Treatment; Saccharomyces Boulardii - During Treatment; Saccharomyces Boulardii - After Treatment: Saccharomyces boulardii: 250 mg, 3 times daily on an empty stomach for 14 days
Arm/Group | Amoxicillin - Before Treatment | Amoxicillin - During Treatment | Amoxicillin - After Treatment | Control | Trametes Versicolor Extract - Before Treatment | Trametes Versicolor Extract - During Treatment | Trametes Versicolor Extract - After Treatment | Saccharomyces Boulardii - Before Treatment | Saccharomyces Boulardii - During Treatment | Saccharomyces Boulardii - After Treatment
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6 | 6 | 7 | 7 | 7
percentage of bacterial genera in stool
  Faecalibacterium | 22.3 (0) | 20.9 (0) | 18.0 (0) | 25.5 (0) | 12.7 (0) | 22.6 (0) | 12.6 (0) | 19.3 (0) | 25.2 (0) | 21.2 (0)
  Bacteroides | 13.9 (0) | 17.9 (0) | 17.3 (0) | 22.3 (0) | 23.6 (0) | 17.6 (0) | 21.8 (0) | 12.6 (0) | 10.8 (0) | 16.6 (0)
  Roseburia | 12.6 (0) | 6.1 (0) | 10.2 (0) | 9.1 (0) | 8.6 (0) | 11.4 (0) | 15.1 (0) | 7.3 (0) | 6.2 (0) | 7.3 (0)
  Clostridium | 7.9 (0) | 9.9 (0) | 9.4 (0) | 6.4 (0) | 11.3 (0) | 8.0 (0) | 12.1 (0) | 10.6 (0) | 10.9 (0) | 10.5 (0)
  Oscillospira | 10.4 (0) | 6.3 (0) | 7.2 (0) | 5.8 (0) | 7.1 (0) | 7.0 (0) | 7.8 (0) | 2.0 (0) | 2.1 (0) | 2.2 (0)
  Dialister | 8.2 (0) | 2.5 (0) | 8.8 (0) | 9.0 (0) | 6.6 (0) | 7.3 (0) | 5.4 (0) | 12.2 (0) | 14.3 (0) | 11.4 (0)
  Ruminococcus | 5.1 (0) | 3.2 (0) | 4.0 (0) | 3.8 (0) | 6.4 (0) | 6.6 (0) | 4.8 (0) | 3.7 (0) | 5.9 (0) | 5.0 (0)
  Coprococcus | 3.1 (0) | 1.8 (0) | 4.0 (0) | 1.8 (0) | 2.8 (0) | 1.8 (0) | 1.8 (0) | 1.9 (0) | 2.2 (0) | 2.9 (0)
  Prevotella | 1.8 (0) | 3.7 (0) | 4.8 (0) | 2.7 (0) | 0.9 (0) | 0.3 (0) | 0.4 (0) | 2.7 (0) | 1.0 (0) | 1.3 (0)
  Blautia | 2.3 (0) | 1.3 (0) | 1.5 (0) | 1.9 (0) | 2.6 (0) | 2.5 (0) | 4.4 (0) | 1.6 (0) | 1.9 (0) | 2.4 (0)
  Escherichia/shigella | 1.2 (0) | 14.8 (0) | 3.0 (0) | 1.5 (0) | 0.5 (0) | 0.2 (0) | 1.0 (0) | 0.9 (0) | 0.3 (0) | 0.3 (0)
  Phascolarctobacterium | 1.6 (0) | 1.2 (0) | 1.4 (0) | 1.6 (0) | 1.7 (0) | 2.0 (0) | 1.5 (0) | 2.4 (0) | 2.2 (0) | 2.6 (0)
  Alistipes | 1.4 (0) | 1.0 (0) | 1.1 (0) | 1.1 (0) | 0.8 (0) | 1.4 (0) | 1.0 (0) | 0.5 (0) | 0.6 (0) | 1.1 (0)
  Anaerotruncus | 0.6 (0) | 0.4 (0) | 0.6 (0) | 0.9 (0) | 1.4 (0) | 1.6 (0) | 2.0 (0) | 0.8 (0) | 0.8 (0) | 0.6 (0)
  Parabacteroides | 0.7 (0) | 1.1 (0) | 1.8 (0) | 1.1 (0) | 0.7 (0) | 0.5 (0) | 0.4 (0) | 2.5 (0) | 0.5 (0) | 1.0 (0)
  Akkermansia | 0.1 (0) | 0.2 (0) | 0.7 (0) | 1.1 (0) | 2.1 (0) | 0.3 (0) | 1.5 (0) | 0.9 (0) | 0.2 (0) | 0.7 (0)
Statistical Analysis 1: Comparison: Amoxicillin - Before Treatment vs Amoxicillin - During Treatment vs Amoxicillin - After Treatment; Statistical analysis was performed using a variety of computer packages including XLstat, NCSS 2007, "R" and NCSS 2010; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Prebiotic | Probiotic | Antibiotic | Control
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 0/8 | 2/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prebiotic (N=8) | Probiotic (N=8) | Antibiotic (N=8) | Control (N=8)
Soft stool (Gastrointestinal disorders) | 0 | 0 | 2 | 0
gas (Gastrointestinal disorders) | 1 | 0 | 0 | 0
constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes